CLINICAL TRIAL: NCT05278234
Title: An Efficacy Trial of Community Health Worker-Delivered Chronic Pain Self-Management Support for Vulnerable Older Adults
Brief Title: STEPS: An Efficacy Trial of a Chronic Pain Self-Management Program for Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Mary Janevic, Associate Research Scientist, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00206235; 1R01AG071511 (NIH)
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants will engage in a 7-week multicomponent chronic pain self-management program.
  Interventions: Behavioral: STEPS
- Usual care control arm (No Intervention): After completing the 12 month telephone survey, control group participants will be given access to the online program, a wearable physical activity tracker to use and keep, and will be invited to attend a workshop that provides key intervention content and individualized goal-setting guidance.

INTERVENTIONS:
Behavioral: STEPS — Participants will initially meet with a community health worker (CHW) for a 1-hour orientation at the participant's home, a Henry Ford Health System site or the University of Michigan Detroit Center, or virtual. The CHW will show participants how to use the web modules. Participants will be given (or mailed) a wearable activity tracker to use throughout the course of the 7-week program. Each week participants will watch a brief video on the STEPS website; they may also be asked to complete handouts in the workbook. They will have a weekly 30-minute telephone session with the CHW. CHWs will review the weekly topic, help participants practice new skills, and set a related goal. CHWs will screen for social needs and make appropriate community referrals. Participants will set walking goals each week, using step-count data from the physical activity tracker. Participants will track daily step counts.
  Other Names: Seniors using Technology to Engage in Pain Self-management
  Arms: Intervention arm

SUMMARY:
The goal of this study is to determine whether community health workers (CHWs)-i.e., lay health workers with close ties to the communities they serve - can effectively teach cognitive-behavioral pain management strategies to older adults in a disadvantaged urban setting. Specific aims are: to test, in a sample of 414 primarily African American older adults, whether the STEPS pain self-management intervention, delivered over 7 weeks through telephone sessions with a CHW and mobile health tools, improves pain outcomes at 2 and 12 months compared to a usual care control group. We will also assess the mechanisms by which the intervention may bring about positive changes in pain outcomes. We will use mixed quantitative and qualitative methods to assess participant engagement and satisfaction, and factors affecting implementation.

ELIGIBILITY:
Inclusion Criteria:

* Community-living
* Have a cell or landline phone
* Self-reported chronic musculoskeletal pain (pain in muscles or joints for >= 3 months); >=4 (0-10 scale) average pain level over last week; >=1 day/previous 30 when pain made it difficult to do usual activities.
* Able to converse comfortably in English

Exclusion Criteria:

* Serious acute illness or hospitalization in last month
* Planned major surgery in next three months that would interfere with program participation (e.g., knee or hip replacement);
* Severe cognitive impairment or other severe physical or psychiatric disorder judged by study team to pose significant barrier to participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Interference | Baseline, 2 months from baseline, and 12 months from baseline
  The Pain Interference 6-item subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-43 Adult Profile. Items ask how much pain in the last 7 days has interfered with daily activities such as household chores and social activities (1=not at all to 5=very much); raw total scale scores range from 6 (low interference) to 30 (high interference). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 42 to 76, with a higher score representing worse outcome.

SECONDARY OUTCOMES:
Participant Global Impression of Change--Pain | 2 months from baseline, and 12 months from baseline
  How participant thinks their pain has changed from baseline (much worse (1) to much better (7)). Higher score represents a better outcome.
Participant Global Impression of Change - Functioning | 2 months from baseline, and 12 months from baseline
  How participant thinks their functioning has changed from baseline (much worse (1) to much better (7)). Higher score represents a better outcome.
Change in pain intensity | Baseline, 2 months from baseline, and 12 months from baseline
  A numeric rating scale ranging from 0 (no pain at all; best outcome) to 10 (worst pain you can imagine; worst outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Janevic MR, Lindsay R, Brines E, Wisdom K, Robinson-Lane SG, Brewer R, Murphy SL, Piette J, Grijalva L, Anderson M, Clement J, Latimer C. A community health worker-delivered intervention (STEPS) to support chronic pain self-management among older adults in an underserved urban community: protocol for a randomized trial. Trials. 2025 Jun 2;26(1):186. doi: 10.1186/s13063-025-08892-w. PMID 40457457

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT05278234/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT05278234/ICF_001.pdf